CLINICAL TRIAL: NCT05945537
Title: A Phase 1 Randomised, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of INI-822 in Healthy Volunteers and Participants with Non-alcoholic Steatohepatitis (NASH) or Presumed NASH
Brief Title: A Study of INI-822 in Healthy Volunteers and Participants with Non-alcoholic Steatohepatitis (NASH) or Presumed NASH
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Inipharm Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INI-822-001
Record Dates: First submitted 2023-06-27; First posted 2023-07-14 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (INI-822) (Experimental): Participants will receive INI-822 orally once daily.
  Interventions: Drug: INI-822 (A)
- B (Placebo) (Placebo Comparator): Participants will receive placebo orally once daily.
  Interventions: Other: Placebo (B)

INTERVENTIONS:
Drug: INI-822 (A) — Different dose levels of INI-822
  Arms: A (INI-822)
Other: Placebo (B) — Matching placebo to INI-822
  Arms: B (Placebo)

SUMMARY:
This Phase 1 trial will explore the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single and multiple ascending doses of INI-822 in healthy volunteers in Parts A, B, and D and in participants with a history of NASH or presumed NASH in Part C.

DETAILED DESCRIPTION:
The study will consist of 4 parts:

Approximately 104 participants are planned to be enroled into the study.

* In Part A (SAD), approximately 48 healthy adult participants are planned to be enroled in 6 cohorts of 8 participants each (Cohorts A1 to A6, including one fasted:fed crossover cohort to assess food effect).
* In Part B (MAD), approximately 24 healthy adult participants are planned to be enroled in 3 cohorts of 8 participants each (Cohorts B1 to B3).
* In Part C (Pharmacodynamics), approximately 24 participants with NASH or presumed NASH are planned to be enroled in 2 cohorts of 12 participants each (Cohorts C1 to C2).
* In Part D (SAD), approximately 8 healthy adult participants are planned to be enroled in 1 Cohort of 8 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Females must not be pregnant or lactating, and must use acceptable, highly effective double contraception (see Section 7.3.1) from Screening until 90 days after their last dose of IP or 5 half-lives, whichever is longer. Females with same-sex partners (abstinent from penile-vaginal intercourse) or who are abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and Day -1. Women not of childbearing potential must be postmenopausal for ≥ 12 months (postmenopausal status is to be confirmed through testing of follicle stimulating hormone [FSH] levels ≥ 40 IU/L at Screening for amenorrhoeic female participants). Females must not donate ova from the first dose of IP until at least 90 days after the last dose of IP or 5 half-lives, whichever is longer.
2. Males must be surgically sterile (> 30 days since vasectomy [documented evidence] with no viable sperm), or, if engaged in sexual relations with a WOCBP, they must use a condom and either his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or an acceptable, highly effective contraceptive method (see Section 7.3.1) must be used from Day -1 until study completion. Males with same-sex partners (abstinent from penile-vaginal intercourse) or abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle. males must not donate sperm from the first dose of IP until at least 90 days after the last dose of IP or 5 half-lives, whichever is longer.
3. Able and willing to attend the necessary visits to the study site.
4. Able and willing to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.
5. Normal renal function (estimated glomerular filtration rate > 60 mL/min using Cockcroft-Gault).

   For Parts A and B only:
6. Clinical laboratory values within normal range at Screening and Day -1 and Day 7 (Part D), as specified by the testing laboratory, unless deemed not clinically significant by the Investigator or designee. Any laboratory values > upper limit of normal (ULN) at Screening should be discussed with the Sponsor, independent Medical Monitor (MM), or Investigator for approval prior to inclusion. Repeat testing at Screening is acceptable for out-of-range values following approval by the Investigator or designee. Inclusion of participants with laboratory values > ULN at Day -1 and Day 7 (Part D) will be at the Investigator's discretion.
7. In good general health, with no significant medical history, and no clinically significant abnormalities on physical examination at Screening and/or before the first administration of IP, at the discretion of the Investigator or designee.
8. Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2 with a maximum body weight of 120 kg.
9. 18 to 55 years of age (inclusive at the time of informed consent).
10. Able and willing to refrain from use of tobacco and other nicotine-containing products while at the study site and through the study treatment period.

For Part C only:

11.18 to 65 years of age (inclusive at the time of informed consent).

12. A diagnosis of NASH confirmed by 1 or more of the following:

1. Historical liver biopsy consistent with NASH (presence of Grade 1 steatosis, hepatocellular ballooning, and lobular inflammation) according to the non-alcoholic fatty liver disease (NAFLD) activity score.
2. F0-3 fibrosis according to the NASH Clinical Research Network classification within 1 year of Screening.
3. A clinical diagnosis of NASH, and the presence of any component of the metabolic syndrome (obesity, dyslipidemia, hypertension, elevated fasting glucose, or type 2 diabetes).
4. FibroScan-aspartate aminotransferase (FAST) score more than equal to 0.35.

   13. Alanine aminotransferase (ALT) > 1.00 × ULN at 2 separate time points in the past 6 months. At least 1 time point must be at Screening and the values must be at least 2 weeks apart. Patients with ALT values <1.00 × ULN may be included in the study on a case-by-case basis after approval by the Sponsor.

   14. Fibrosis-4 (FIB-4) score ≤ 2.67, controlled attenuation parameter (CAP) score by FibroScan® ≥ 280 Db/m, and liver stiffness measurement (LSM) by FibroScan® ≤ 14 kPa.

   15. No documented weight loss > 5% in the 6 months preceding Screening.

   16. If on glucagon-like peptide 1 (GLP1) agonists, sodium-glucose co-transporter 2 (SGLT2) inhibitors, or vitamin E (dose > 400 IU/day), then should have been on a stable dose for at least 3 months.

   17. Platelet count > 150,000 and albumin ≥ 35 g/L.

   18. BMI ≥ 18.0 and ≤ 40.0 kg/m2

Exclusion Criteria:

A participant who meets any of the following exclusion criteria must be excluded from the study:

1. An underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely for the participant to comply with the protocol or complete the study per protocol.
2. Blood donation or significant blood loss (> 500 mL) within 60 days prior to the first administration of IP.
3. Plasma donation within 7 days prior to the first administration of IP.
4. Fever (body temperature > 37.7°C) or symptomatic viral or bacterial infection within 2 weeks prior to Day 1.
5. Dysphagia that would limit ability to swallow IP.
6. History of severe allergic or anaphylactic reactions, or sensitivity to the IP or its constituents. The excipients in the IP are: Hydroxypropylmethylcellulose Acetate Succinate (HPMCAS), Microcrystalline Cellulose, Micronized Poloxamer 407 (polyoxyethylene oxide), Croscarmellose Sodium, Silicon Dioxide, Magnesium Stearate, and Hydroxypropylmethylcellulose capsules containing Titanium Oxide.
7. Abnormalities in physical examination at Screening and Day -1 which are deemed clinically significant by the Investigator or designee.
8. Abnormal electrocardiogram (ECG) measurements at Screening (an average of 3 readings) and Day -1 (single reading) that are considered by the Investigator or designee to be clinically significant, including corrected QT interval with Fridericia's correction (QTcF) > 450 msec (males) or > 470 msec (females).
9. Unstable vital sign(s) or the following values seen at Screening or prior to dosing following 5 minutes of resting in the semi-supine position (an abnormal value may be repeated once, separated by at least 5 minutes, with both values documented):

   1. Systolic blood pressure < 90 mmHg or > 160 mmHg OR
   2. Diastolic blood pressure < 50 mmHg or > 95 mmHg OR
   3. Pulse rate < 45 beats per minute (bpm) or > 100 bpm.
10. History or presence of other causes of liver disease including genetic, autoimmune, viral, and alcoholic liver disease.
11. Cirrhosis of the liver as defined by:

    1. A prior history of decompensated liver disease, including ascites, hepatic encephalopathy, or variceal bleeding OR
    2. F4 on previous liver biopsy OR
    3. Historical evidence of cirrhosis on liver imaging.
12. History of major hospitalisation or major surgery within 6 months prior to Screening. Sites are encouraged to confirm with the Sponsor or Medical Monitor if there are any questions on what would be considered major hospitalization or major surgery.
13. Infections requiring parenteral antibiotics within 6 months prior to Screening.
14. Vaccination with a live vaccine within 4 weeks prior to the first administration of IP.
15. Exposure to any significantly immune suppressing drug (including experimental therapies as part of a clinical study) within 4 months prior to Screening or 5-half lives, whichever is longer.
16. Positive blood screen for active infections including human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) at Screening.
17. History of substance abuse or dependency or history of recreational intravenous drug use over the last 12 months (by self-declaration).
18. Use of any IP or investigational medical device within 30 days for small molecules (or 5 half lives of the IP if longer than 30 days) or 90 days for biologics prior to first IP administration.
19. Anything that the Investigator considers would jeopardise the safety of the participant, prevent complete participation in the study, or compromise interpretation of study data.
20. Bariatric surgery.
21. Cardiovascular disease including heart failure with reduced left ventricular ejection fraction, atrial fibrillation requiring anticoagulation, or any other cardiovascular illness that, in the opinion of the Investigator, warrants exclusion from the study.

    For Parts A and B only:
22. Use of (or anticipated use of) any prescription drugs (other than hormonal contraception; oral contraceptive pills [OCPs], long-acting implantable hormones, injectable hormones, or an intrauterine device [IUD]), any known drugs or supplements that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) enzymes, over-the-counter (OTC) medication, herbal remedies, supplements or vitamins within 48 hours of IP administration and during the course of the study without prior approval of the Investigator and independent MM. Simple analgesia (paracetamol < 2 g/day) may be permitted at the discretion of the Investigator.
23. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, haematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity, as determined by the Investigator.
24. History of or suspected malignancy. Participants with basal or squamous cell carcinoma of the skin or carcinoma in situ that has been successfully treated could be included at the discretion of the Investigator or designee.
25. Positive toxicology screening panel (urine test including Methamphetamine, Opiates, Cocaine, tetrahydrocannabinol, Phencyclidine, Benzodiazepines, Barbiturates, Methadone, tricyclic antidepressants and Amphetamine), or alcohol breath test at Screening or Day -1
26. History of alcohol use disorder (within 9 months prior to Screening by self-declaration) or habitual consumption of significant amounts of alcohol (by self-declaration), defined as > 10 standard drinks per week or > 4 standard drinks on any single day (where 1 standard drink = 360 mL of beer, 45 mL of 40% spirit, or a 150 mL glass of wine). Participants who are unable to abstain from alcohol 72 hours prior to Screening and Day -1 visits and until study completion are to be excluded.

    For Part C only:
27. ALT ≥ 5 × ULN; AST>ALT. If ALT ≤ ULN, then AST may be greater than the ALT if it is also ≤ ULN.
28. Use of (or anticipated use of) any known drugs or supplements that are moderate or strong inhibitors/inducers of CYP enzymes or any drugs that are substrates of CYP2C9 with a narrow therapeutic index (e.g., warfarin or other coumarin based anticoagulants, phenytoin, celecoxib, glimepiride, tolbutamide or phenobarbital or other drugs metabolised by CYP2C9) or any oral drugs that are significantly metabolised by CYP3A4 (e.g., alfentanil, apixaban, avanafil, buspirone, cyclosporine, dihydroergotamine, ergotamine, fentanyl, oxybutinin, losartan, lomitapide, lovastatin, midazolam, naloxegol, nisoldipine, pimozide, quinidine, sildenafil, simvastatin, sirolimus, tadalafil, tamsulosin, tacrolimus and zopiclone), during the course of the study. Prescription medications for stable medical condition may be allowable if the Investigator considers they will not interfere with the study; the independent MM may be contacted to discuss any particular medications.
29. Participants with uncontrolled medical conditions; the independent MM may be contacted for discussion.
30. History of significant cardiovascular disease, including cardiac failure, myocardial infarction, unstable angina, stroke or transient ischaemic attack within 6 months prior to the first dose of IP.
31. Uncontrolled diabetes mellitus (haemoglobin A1c [HbA1c] > 9.0% at Screening).
32. Malignancy within the last 5 years; basal or squamous cell carcinoma of the skin or carcinoma in situ that has been successfully treated could be included at the discretion of Investigator or designee.
33. History or presence of a condition associated with significant immunosuppression.
34. Positive toxicology screening panel (urine test including Methamphetamine, Opiates, Cocaine, tetrahydrocannabinol, Phencyclidine, Benzodiazepines, Barbiturates, Methadone, and Amphetamine) at Screening or Day -1. A positive toxicology screening that is explained by a prescribed medication is allowable.
35. History of alcohol use disorder (within 9 months prior to Screening by self-declaration) or habitual consumption of significant amounts of alcohol (by self-declaration), defined as > 10 standard drinks per week or > 4 standard drinks in a day (where 1 standard drink = 360 mL of beer, 45 mL of 40% spirit, or a 150 mL glass of wine). Participants who are unable to abstain from alcohol 72 hours prior to Screening and Day -1 visits are to be excluded. Participants unable to consume 10 standard drinks or fewer in a week or 2 standard drinks in a day or fewer during the study are to be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs). | Part A: Up to 5 Weeks
  AEs will be graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Incidence of adverse events (AEs). | Part A fasted fed crossover cohort: Up to 8 weeks
  AEs will be graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Incidence of adverse events (AEs). | Part B: Up to 7 weeks
  AEs will be graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Incidence of adverse events (AEs). | Part C: Up to 9 weeks
  AEs will be graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of participants with clinical laboratory abnormalities | Part A: Up to 5 Weeks
Number of participants with clinical laboratory abnormalities | Part A fasted fed crossover cohort: Up to 8 weeks
Number of participants with clinical laboratory abnormalities | Part B: Up to 7 weeks
Number of participants with clinical laboratory abnormalities | Part C: Up to 9 weeks

SECONDARY OUTCOMES:
Plasma area under the curve (AUC) from time 0 to t (AUC0-t) | Part A: Up to 5 Weeks, Part A fasted fed crossover cohort: Up to 8 weeks, Part B: Up to 7 weeks, Part C: Up to 9 weeks
AUC from time 0 to infinity (AUC0-inf) | Part A: Up to 5 Weeks, Part A fasted fed crossover cohort: Up to 8 weeks, Part B: Up to 7 weeks, Part C: Up to 9 weeks
Maximum concentration (Cmax) | Part A: Up to 5 Weeks, Part A fasted fed crossover cohort: Up to 8 weeks, Part B: Up to 7 weeks, Part C: Up to 9 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (7):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - CMAX Clinical Research, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria